CLINICAL TRIAL: NCT03302312
Title: A Randomized, Sham-procedure-controlled, Blinded Study to Evaluate the Effectiveness and Acceptability of Right-sided Stellate Ganglion Block for Treatment of Posttraumatic Stress Disorder Symptoms - Acceptability
Brief Title: Effectiveness and Acceptability of Stellate Ganglion Block for Posttraumatic Stress Disorder Symptoms - Acceptability
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Collaborators: Womack Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency); Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SGB-201a
Record Dates: First submitted 2017-09-28; First posted 2017-10-05 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Generalized Anxiety Disorder; Depression; Distress; Alcohol Use; Pain
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Depression; Alcohol Drinking; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants: Service members who received at least one SGB study procedure as part of the clinical effectiveness trial during the three months prior to qualitative data collection or service members who received at least one SGB for PTSD symptoms at a study site in the three months prior to qualitative data collection.
- Providers: Behavioral Health or other (e.g., Family Medicine) clinicians who have referred or could potentially have referred service members for SGB for PTSD symptoms, as well as physicians who provide SGBs.

SUMMARY:
This qualitative study will use focus groups, small group interviews, and individual interviews (both in person and over the phone) to compile a range of perspectives on service members' decision-making processes and information needs related to Stellate Ganglion Block (SGB). Participants will include service members, spouses, and providers.

DETAILED DESCRIPTION:
The qualitative (acceptability) study will use focus groups, small group interviews, and individual interviews (both in person and telephonic) to compile a range of perspectives on service members' decision-making processes and information needs related to SGB. Participants will include service members, spouses, and providers. Data collection will occur at each study site because attitudes conveyed by leadership and chain of command may vary across installation. Scheduling will be based on the accumulation of ample service members indicating an interest in participating.

All service members enrolled in the clinical effectiveness trial (Study Number: NCT03077919) will be eligible for the qualitative study if they have received at least one SGB study procedure during the three months prior to qualitative data collection. When qualitative data collection is scheduled, the study team will approach service members who indicated initial interest in participating in the acceptability if they still meet the eligibility criteria. Service members will not be contacted for qualitative study participation if the Research Coordinator or treating provider considers that participation would cause undue distress based on their most recent contact with the individual.

Service members who did not participate in the clinical effectiveness trial are eligible for the qualitative study if they have received at least one SGB for PTSD symptoms at a study site in the three months prior to qualitative data collection and if participation would not cause undue distress. These participants will be recruited in the clinic as well as through a medical record search conducted by the Site PI or other clinical staff.

Assignment to specific focus groups will be based on pay grade and subjective assessment of change as reported at the 4-Week assessment or at the time of screening for the qualitative study. In order to maximize homogeneity, lower enlisted service members and non-commissioned officers (NCOs) will be assigned to different groups. These groups will be further divided so that those reporting positive change since the procedure will be assigned to a different group than those reporting no change or feeling worse than at the time of the procedure. Depending on the number of eligible participants by pay grade, officers may be interviewed individually.

Eligible service members, both clinical trial and non-clinical trial participants, may be assigned to a service member/spouse dyad subgroup if they meet the above criteria and their spouse has expressed an interest in participating in the qualitative study. Those service members who participate as part of the dyad subgroup will not be eligible to participate in the service member only focus groups.

Eligible participants for the provider focus groups will be Behavioral Health or other (e.g., Family Medicine) clinicians who have referred or could potentially refer service members for SGB for PTSD symptoms, as well as physicians who provide SGBs.

The planned focus group interviews will be structured discussions on a particular topic involving a small number of people under the direction of a moderator (Krueger & Casey, 2000). The method relies on both the interactive social context of the discussion and on the individual experiences of each of the group members to produce a rich discussion in which shared experiences stimulate individual contributions.

The qualitative study will explore participants' perceptions of SGB in relation to other options for treatment of PTSD, from the perspectives of service members, service member/spouse couples, and providers. Broad topics covered in service member focus groups, service members/spouse interviews, and provider focus group are:

* Context for mental health and treatment
* Advantages and drawbacks of treatment options
* Information and decision-making
* Experience and expectations

Focus groups and small group interviews will take approximately 90 minutes, service member-significant other interviews will take approximately 60 minutes, and individual interviews will take approximately 45 minutes.

All focus groups and interviews will be led by a study team member with prior experience in qualitative data collection with clinicians and service members engaged in mental health treatment. Real-time notes will be collected by a second team member but each focus group or interview will also be audio-recorded if all participants give permission to do so. The purpose of the audio recordings is to augment any notes taken by the second team member.

Data from focus groups and interviews will be summarized in topline notes as soon as feasible after data collection. In-depth analysis will employ standard qualitative methods. All notes will be entered into qualitative data base software such as NVivo 9 (QSR International Pty Ltd. Version 9, 2010) to facilitate coding and retrieval. Analysis will be both deductive, following a hierarchical coding structure based on topic guide questions, and inductive, creating queries to assess patterns observed in the data and hypotheses emerging from preliminary analyses. Analytical matrixes to compare responses across respondent types will also be constructed. Comparisons of interest include enlisted, NCO, officer; service member, spouse; service member, provider; self-assessed improvement, no self-assessed improvement; Behavioral Health clinicians, Family Medicine physicians; and study sites

ELIGIBILITY:
Inclusion criteria:

* Service members must have received at least one SGB and/or study procedure for PTSD symptoms during the past three months at a participating study site (as a participant in the clinical effectiveness trial or outside of the study).
* Clinical trial participants must have indicated willingness to participate in the qualitative study when asked by the Research Coordinator (RC) at baseline data collection.
* Non-clinical trial participants must be active-duty status.
* A service member/spouse dyad will consist of a service member meeting an above criterion and his/her spouse.
* Providers will be Behavioral Health or other (e.g., Family Medicine) clinicians who have referred or could potentially have referred service members to the study, and physicians who administer SGBs.

Exclusion Criteria:

• Service members will be excluded from the qualitative study if participation would cause them undue distress, in the opinion of the RC or treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * participants in effectiveness clinical trial and their spouses
  * service members who have received SGB for PTSD symptoms at the participating study sites outside of the clinical trial and their spouse
  * providers who have referred or could potentially have referred patients for SGB for PTSD symptoms at the study sites
  * clinicians who provide SGB for PTSD
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Participants' perceptions of SGB in relation to other options for treatment of PTSD, from the perspectives of service members or service member/spouse couples. | Within three month of receiving one SGB study procedure for PTSD symptoms
  Discussion topic areas:
  * Context for mental health and treatment
  * Advantages and drawbacks of treatment options
  * Information and decision-making
  * Experience and expectations
Participants' perceptions of SGB in relation to other options for treatment of PTSD, from the perspectives of providers | Through study completion, approximately six months
  Discussion topic areas:
  * Context for mental health and treatment
  * Advantages and drawbacks of treatment options
  * Information and decision-making
  * Experience and expectations

CONTACTS AND LOCATIONS:
Overall Officials: Bradford B Walters, MD, PhD, MBA, Principal Investigator — RTI International
Locations (3):
- United States (2):
  - Tripler Army Medical Center (TAMC), Honolulu, Hawaii
  - Womack Army Medical Center (WAMC), Fort Bragg, North Carolina
- Landstuhl Regional Medical Center (LRMC), Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krueger, R.A., & M.A. Casey, M. A. (2000). Focus groups. A practical guide for applied research. Thousand Oaks, CA: Sage.